CLINICAL TRIAL: NCT03559179
Title: Clinical Decision Support for Opioid Use Disorders in Medical Settings: Pilot Usability Testing in an EMR
Brief Title: Clinical Decision Support for Opioid Use Disorders in Medical Settings: Usability Testing in an EMR
Acronym: COMPUTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0076-ot; 3UG1DA040316-03S1 (NIH)
Record Dates: First submitted 2018-05-09; First posted 2018-06-18 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2019-02

CONDITIONS: Opioid-use Disorder
Keywords: CDS; Medication Assisted Therapy
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waivered Providers Receive the Opioid Wizard (Experimental): All providers who have a buprenorphine waiver will receive the OUD clinical decision support tool (Opioid Wizard).
  Interventions: Other: Opioid Wizard
- Does not Receive the Opioid Wizard (No Intervention): All non-buprenorphine waivered providers will be randomized to receive or not receive the Opioid Wizard. This arm of providers will continue to treat their patients as usual.
- Non-Waivered Providers who receive Opioid Wizard (Experimental): All non-buprenorphine waivered providers will be randomized to receive or not receive the Opioid. This arm of providers will receive the OUD clinical decision support tool (Opioid Wizard).
  Interventions: Other: Opioid Wizard

INTERVENTIONS:
Other: Opioid Wizard — The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
  Arms: Non-Waivered Providers who receive Opioid Wizard; Waivered Providers Receive the Opioid Wizard

SUMMARY:
The primary objective of this pilot study is to program an opioid use disorder (OUD) clinical decision support (CDS) tool for use in an electronic medical record (EMR) and obtain high primary care physician (PCP) usability and acceptability. The OUD-CDS is based on the NIDA-Blending Initiative white paper, "Clinical Decision Support for Opioid Use Disorders: Working Group Report," which itself is based on national evidence-based guidelines (American Society of Addiction Medicine (ASAM 2015), VA (VA 2015). As such, this pilot study aims to help PCPs achieve accepted standards of care in OUD treatment. The secondary objectives of this pilot study are to evaluate the usefulness of the tool by comparing OUD case-finding, medication-assisted therapy (MAT) and referral patterns pre- and post-CDS deployment for PCPs with and without CDS access.

ELIGIBILITY:
Inclusion Criteria:

* Be an MD, Doctor of Osteopathy, Nurse Practitioner or Physician's Assistant engaged in independent primary care of adults at HealthPartners or Park Nicollet
* Have at least schedule 3 DEA prescribing privileges
* Voluntarily provide written informed consent to participate in this study

Exclusion Criteria:

* Less than half-time clinical primary care responsibilities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Rossom RC, Sperl-Hillen JM, O'Connor PJ, Crain AL, Nightingale L, Pylkas A, Huntley KV, Bart G. A pilot study of the functionality and clinician acceptance of a clinical decision support tool to improve primary care of opioid use disorder. Addict Sci Clin Pract. 2021 Jun 15;16(1):37. doi: 10.1186/s13722-021-00245-7. PMID 34130758

RESULTS

PARTICIPANT FLOW:
Groups:
- Waivered Providers Received the Opioid Wizard: All Buprenorphine-Waivered providers received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Non-Waivered Providers Received The Opioid Wizard: Non-buprenorphine waivered providers were randomized to receive/not receive the Opioid Wizard. This arm represents providers who received the Opioid Wizard.
- Non-Waivered Providers Who Did Not Receive the Opioid Wizard: Non-Buprenorphine waivered providers are randomized to receive/not receive the Opioid Wizard. This arm represents providers who did not receive the Opioid Wizard. These providers continued to treat their patients as usual.
Period: Overall Study
Arm/Group | Waivered Providers Received the Opioid Wizard | Non-Waivered Providers Received The Opioid Wizard | Non-Waivered Providers Who Did Not Receive the Opioid Wizard
Started | 8 | 24 | 23
Completed | 8 | 23 | 23
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Waivered Providers Received the Opioid Wizard: These providers received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Non-Waivered Providers Who Received the Opioid Wizard: Non-Buprenorphine waivered providers were randomized to receive/not receive the Opioid Wizard. This arm represents non-waivered providers who received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Non-Waivered Providers Who do Not Receive the Opioid Wizard: These are non-buprenorphine waivered providers continued to treat their patients as usual.
- Total: Total of all reporting groups
Arm/Group | Waivered Providers Received the Opioid Wizard | Non-Waivered Providers Who Received the Opioid Wizard | Non-Waivered Providers Who do Not Receive the Opioid Wizard | Total
Number analyzed (Participants) | 8 | 24 | 23 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 23 | 23 | 54
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 16 | 33
  Male | 4 | 11 | 7 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 19 | 18 | 42
  Black | 1 | 1 | 1 | 3
  Asian | 0 | 4 | 2 | 6
  Multiple | 1 | 0 | 1 | 2
  Unknown | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intervention PCP Confidence in Assessing and Treating OUD
Description: # of intervention PCPs who report feeling "moderately" or "very" confident in assessing and treating OUD.
Time Frame: This outcome measure was calculated at approximately month 10 of the pilot study
Population: This outcome was to help show proof of the OUD-CDS concept using responses from intervention PCPs. One intervention provider stopped working for the organization during the intervention. Two additional intervention providers in the "Non-Waivered providers who received the Opioid Wizard" arm did not complete follow-up surveys.
Measure: Count of Participants; unit: Participants
Groups:
- Non-Waivered Providers Who Received the Opioid Wizard: Non-Buprenorphine waivered providers were randomized to receive/not receive the Opioid Wizard. This arm represents providers who received the Opioid Wizard.
Arm/Group | Waivered Providers Received the Opioid Wizard | Non-Waivered Providers Who Received the Opioid Wizard
Number analyzed (Participants) | 8 | 21
Participants
  # of INT PCPs reporting confidence assessing OUD | 6 | 11
  # of INT PCPs reporting confidence treating OUD | 8 | 1

2. Primary Outcome: Intervention PCP Likeliness to Recommend Use of the OUD-CDS
Description: # of PCPs with CDS access who rate the OUD-CDS >4 on a 5-point Likert scale of likeliness to recommend use of the tool to their colleagues. The scale ranges from 1-"not at all likely" to 5-"very likely," with higher values representing a higher likelihood of recommending the OUD-CDS to other colleagues.
Time Frame: This was calculated after PCP surveys were completed, approximately month 10
Population: One non-waivered intervention provider stopped working for the organization and two additional non-waivered intervention providers did not complete the follow-up survey.
Measure: Count of Participants; unit: Participants
Groups:
- Waivered Providers Receive the Opioid Wizard: All providers who have a buprenorphine waiver received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Non-Waivered Providers Who Receive Opioid Wizard: All non-buprenorphine waivered providers were randomized to receive or not receive the Opioid. This arm of providers received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
Arm/Group | Waivered Providers Receive the Opioid Wizard | Non-Waivered Providers Who Receive Opioid Wizard
Number analyzed (Participants) | 8 | 21
Participants | 6 | 13

3. Secondary Outcome: Compare Pre- and Post-intervention Rates of OUD Diagnosis in High-risk Patients.
Description: Calculate and compare the number of patients diagnosed with OUD pre- and post-intervention. This will be presented as rate of OUD diagnoses per patient year.
Time Frame: This was calculated at the end of the pilot study (month 8).
Measure: Number; unit: OUD diagnosis per patient year
Groups:
- Waivered Providers Received the Opioid Wizard: All providers who have a buprenorphine waiver received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Non-Waivered Providers Who Received Opioid Wizard: All non-buprenorphine waivered providers were randomized to receive or not receive the Opioid. This arm of providers received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Did Not Receive the Opioid Wizard: All non-buprenorphine waivered providers were randomized to receive or not receive the Opioid Wizard. This arm of providers continued to treat their patients as usual.
Arm/Group | Waivered Providers Received the Opioid Wizard | Non-Waivered Providers Who Received Opioid Wizard | Did Not Receive the Opioid Wizard
Number analyzed (Participants) | 8 | 24 | 23
OUD diagnosis per patient year | 11.3 | 28.54 | 7.87

4. Secondary Outcome: Compare Pre- and Post-intervention Rates of Medication-assisted Therapy (MAT) Use.
Description: Calculate and compare the rate of MAT use among patients with OUD pre- and post-intervention. This is presented as a pre/post ratio of MAT rx per patient year.
Time Frame: This was calculated at the end of the pilot study (month 8).
Measure: Number; unit: pre/post ratio MAT Rx per patient year
Groups:
- Non-Waivered Providers Who Receive the Opioid Wizard: Non-Buprenorphine waivered providers were randomized to receive/not receive the Opioid Wizard. This arm represents non-waivered providers who received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
Arm/Group | Waivered Providers Received the Opioid Wizard | Non-Waivered Providers Who Receive the Opioid Wizard | Non-Waivered Providers Who do Not Receive the Opioid Wizard
Number analyzed (Participants) | 8 | 24 | 23
pre/post ratio MAT Rx per patient year | 1.4 | 1.1 | 1.03

5. Secondary Outcome: Compare Post-intervention Referral Patterns Between Intervention and Control Groups
Description: Calculate and compare how often patients diagnosed with OUD are referred to specialty care or inpatient treatment post-intervention. Compare these rates between intervention and control groups.
Time Frame: This was calculated at the end of the pilot study (month 8).
Measure: Number; unit: post/pre ratio of referral per pt. year
Groups:
- Non-Waivered Providers Who Did Not Receive the Opioid Wizard: These are non-buprenorphine waivered providers continued to treat their patients as usual.
Arm/Group | Waivered Providers Received the Opioid Wizard | Non-Waivered Providers Who Received the Opioid Wizard | Non-Waivered Providers Who Did Not Receive the Opioid Wizard
Number analyzed (Participants) | 8 | 24 | 23
post/pre ratio of referral per pt. year | 0.99 | 1.21 | 1.04

ADVERSE EVENTS:
Time Frame: These data were collected during the entire active intervention period, from 6/6/2018-12/6/2018
Groups:
- Waivered Providers Who Received the Opioid Wizard: These providers received the OUD clinical decision support tool (Opioid Wizard).
  Opioid Wizard: The Opioid Wizard is an OUD clinical decision support tool for primary care providers.
- Non-Waivered Providers Who Received the Opioid Wizard: Non-waivered providers were randomized to receive/not receive the Opioid Wizard.
  This arm represents the providers who received access to the opioid wizard.
- Non-Waivered Providers Who Did Not Receive the Opioid Wizard: Non-waivered providers were randomized to receive/not receive the Opioid Wizard.
  This arm represents the providers who did not receive access to the opioid wizard.These providers continued to treat their patients as usual.
Arm/Group | Waivered Providers Who Received the Opioid Wizard | Non-Waivered Providers Who Received the Opioid Wizard | Non-Waivered Providers Who Did Not Receive the Opioid Wizard
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/8 | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03559179/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03559179/SAP_002.pdf
  • Informed Consent Form (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/79/NCT03559179/ICF_003.pdf